CLINICAL TRIAL: NCT04816994
Title: Effect of Cannabis Extract on Acute Radicular Pain and on Analgesic Requirement: A Double Blinded, Randomized, 24 Hours Follow-up Study
Brief Title: Effect of Cannabis Extract on Acute Radicular Pain and on Analgesic Requirement
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 0092-17-HMO
Record Dates: First submitted 2021-02-08; First posted 2021-03-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Acute Radicular Back Pain; Cannabis
Keywords: Acute radicular back pain; Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High dose cannabis oil (Experimental): Single-dose 20.0 mg tetrahydrocannabinol + 20 mg cannabidiol, Sub-linguistic.
  Interventions: Drug: Single-dose of cannabis oil
- Low dose cannabis oil (Experimental): Single-dose 10 mg tetrahydrocannabinol + 10 mg cannabidiol, Sub-linguistic.
  Interventions: Drug: Single-dose of cannabis oil
- Control (Placebo Comparator): Single-dose Olive oil that is similar in appearance and taste to cannabis oil
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Single-dose of cannabis oil — Single-dose of cannabis oil in order to treat acute radicular pain
  Arms: High dose cannabis oil; Low dose cannabis oil
Drug: Control — Giving a sub-linguistic olive oil that is similar in appearance and taste to cannabis oil
  Arms: Control

SUMMARY:
Clinical evidence about the effects of cannabis in the management of acute pain is rather scarce, mostly consisting of case report-based opinions on adverse events during or after general anesthesia after smoking cannabis, experimental pain trials in healthy volunteers, and a few clinical trials using different drugs, dosages and routes of administration. It is difficult to draw strong conclusions from the available evidence, that may seem sometimes even contradictory, mainly due -the investigators believe- to the many sources of variability in the study designs (e.g.: heterogeneity of the study samples, underpowered, unblinding, lack of randomization, timing of the therapeutic intervention, different experimental pain models, inclusion of different kind of surgical pain, etc.). Nevertheless, expert's opinion after a critical review of the literature is that cannabis and cannabinoids may have a beneficial role in the management of acute pain, at least for a selected group of patients and through an appropriate therapeutic intervention.

Cannabis oil seem to be most suitable to our investigation. The co-administration of tetrahydrocannabinol (THC) with cannabidiol (CBD) may translate into additional therapeutic benefits with an attenuation of adverse effects. And will help treat acute radicular back pain and for renal colic.

DETAILED DESCRIPTION:
Suitable candidates who meet the inclusion criteria will be approached to participate.

Patients hospitalized with a diagnosis of acute radicular pain or pain due to renal colic in the emergency department of the Hadassah Medical Center - Ein Kerem Hebrew University. The indications for performing the treatment are: strong (sharp) pain that lasts for several days and radiates from the back to the leg (ie radicular pain) or pain due to a renal colic. Patients that are suffering from severe enough pain that drives them to the emergency room. The study focuses on patients suffering from radiating nerve pain on the background of acute dyskopia = pain resulting from pressure and inflammation on a nerve root causing sciatic pain and also on patients suffering from renal colic.

This study aims to evaluate the efficacy of cannabis for the treatment of radicular pain and renal colic pain.

These patients will usually also be treated with opiate-type painkillers due to the intense pain. We will test whether there is pain relief and a reduction in the need to use opiates. After oral and written informed consent has been obtained, all patients will be admitted for observational treatment as is customary for a pain patient connected to a PCA pump for 24 hours. After Administering an initial loading dose of morphine 0.05-0.1 mg/kg intravenously, as is customary in a pain patient, the patient will be connected to an accepted protocol of morphine infusion for pain relief under the patient's control as follows: 1 mg upon request, 10 minutes downtime, no background , a maximum hourly dose of 6 mg. The patients will be randomly assigned to one of the following dose groups: 1. High dose of cannabis oil: drops of oil to administer under the tongue (21.6 mg THC, 20 mg CBD). 2. High dose of cannabis oil in split form: half a dose at time t0, half a dose an hour later. b oil drops to administer under the tongue (21.6 mg THC, 20 mg CBD). 3. Low dose of cannabis oil: oil drops to administer under the tongue (10.8 mg THC, 10 mg CBD. 4. Placebo control: A control group will receive olive oil, which is similar in taste and appearance to cannabis oil. The treatments will be given so that the subjects, the researchers-therapists and the results analysts will remain blinded until the end of the recruitment. Blinding of the research drug will be obtained by using similar bottles of the cannabis or placebo-olive oil which will be given in a similar container coated with the same cover and with the same taste. In order to maintain blinding even in the split dose, all other groups will receive the placebo after one hour. It should be noted that participants in the study will continue to receive the standard treatment currently given to patients in the same condition

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years
* ASA 1 or 2
* Acute Radicular Pain < 12 weeks
* Pain of VAS 6 or more/ VRS moderate or more
* Radicular pain: Dermatomal pain that corresponds to physical exam and CT/MRI in the last year

Exclusion Criteria:

* Age < 18 or > 70 years
* ASA 3 or more
* Chronic radicular pain > 12 weeks
* Past spine surgery
* Intermittent Claudication due to Vascular Disease
* Diagnosed Diabetic Neuropathy
* Regular Cannabis use in past 6 months (more than once a week) OR once in last 2 weeks
* Regular opioid use in past week (Targin, Percocet, Tramadol) (Equivalent to Oxycodone 20 mg/day or more)
* Pregnancy or Lactating
* Ischemic heart disease
* Renal or hepatic failure
* History of psychiatric illness
* Cognitive impairment or inability to answer questions
* Known allergy to opioids
* Potential Loss to follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
opioid consumption via - Patient controlled administration (PCA) | The change over 24 hours
  Count of patient-controlled analgesia pushes.

SECONDARY OUTCOMES:
Nausea and vomiting (PONV) score | The change over 24 hours
  PONV score (0 - 4). Before administering baseline, after 0.5, 1, 2, 4, 8 12, 18, 24 h.
Anxiety - VAS | The change over 24 hours
  Self-assessed anxiety visual analog scale (0-100 mm). Before administering baseline, after 0.5, 1, 2, 4, 8 12, 18, 24 h.
VAS | The change over 24 hours
  Self-reported visual analog scale (VAS 0 - 100 mm) at rest and on movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No